CLINICAL TRIAL: NCT02258360
Title: The Effect of Therapeutic Hypothermia After Cardiac Arrest on the Haemostasis.
Brief Title: Hypothermia and Hemostasis After Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROID7005
Record Dates: First submitted 2014-08-29; First posted 2014-10-07 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Hypothermia; Heart Arrest; Hemostasis; Coagulants
Keywords: Thromboelastometry; Haemostasis; Hypothermia; Heart Arrest
MeSH Terms: conditions — Hypothermia; Heart Arrest | interventions — Hypothermia, Induced

ARMS (2):
- 24 hours hypothermia (Active Comparator): Therapeutic hypothermia for 24 hours after reaching target temperature
  Interventions: Other: Therapeutic hypothermia
- 48 hours hypothermia (Experimental): Therapeutic hypothermia for 48 hours after reaching target temperature
  Interventions: Other: Therapeutic hypothermia

INTERVENTIONS:
Other: Therapeutic hypothermia — Therapeutic hypothermia with a target temperature between 32-34°C.

SUMMARY:
This is a sub-study to the Time-differentiated Therapeutic Hypothermia (TTH48, ClinicalTrials.gov Identifier: NCT01689077). TTH48 compares 24 with 48 hours of therapeutic hypothermia at a target temperature of 32-34°C in survivors of out-of-hospital cardiac arrest.

The overall aim of this sub-study is to examine the hemostasis in patients resuscitated after cardiac arrest and treated with 24 and 48 hours of therapeutic hypothermia

Our specific aims are:

* To investigate the whole blood coagulation using the rotational thromboelastometry.
* To investigate the function of platelets

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest of presumed cardiac cause
* Return of spontaneous circulation (ROSC)
* Glasgow Coma Score < 8
* Age > 18 years and < 80 years

Exclusion Criteria:

* > 60 minutes from the circulatory collapse to ROSC
* Time interval > 4 hours from cardiac arrest to initiation of therapeutic hypothermia
* Terminal illness
* Coagulation disorder
* Unwitnessed asystolia
* Cerebral performance category 3-4 before the cardiac arrest
* Severe persistent cardiogenic shock
* Pregnancy
* Persistent cardiogenic shock (systolic blood pressure < 80 despite inotropic treatment)
* New apoplexy or intracerebral hemorrhage
* Lack of consent from the relatives
* Lack of consent from the GP
* Lack of consent from the patient if he/she wakes up and is relevant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clotting time in seconds, EXTEM | After 46 hours
  Measured by thomboelastometry on the ROTEM®
Area under the curve, COL-test | After 46 hours
  Platelet function will be measured using Multiplate®

SECONDARY OUTCOMES:
Clotting time in seconds, EXTEM | After 22 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Clotting time in seconds, -INTEM, FIBTEM and HEPTEM | After 22 hours, 46 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Clot formation time in seconds, -EXTEM, INTEM, FIBTEM and HEPTEM | After 22 hours, 46 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Maximum clot firmness (mm), -EXTEM, INTEM, FIBTEM and HEPTEM | After 22 hours, 46 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Area under the curve, COL-test | After 22 hours and 70 hours
  Platelet function will be measured using Multiplate®.
Area under the curve,- ADP, ASPI and TRAP-test. | After 22 hours, 46 hours and 70 hours
  Platelet function will be measured using Multiplate®.
Time to maximum velocity (s), -EXTEM, INTEM, FIBTEM and HEPTEM | After 22 hours, 46 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Maximum velocity (mm/min), -EXTEM, INTEM, FIBTEM and HEPTEM | After 22 hours, 46 hours and 70 hours
  Measured by thomboelastometry on the ROTEM®.
Area under the curve, Clot stability test | After 22 hours, 46 hours and 70 hours
Area under the curve, Thrombin generation | After 22 hours, 46 hours and 70 hours

OTHER OUTCOMES:
International normalized ratio | After 22 hours, 46 hours and 70 hours
APTT (activated partial thromboplastin time) in seconds | After 22 hours, 46 hours and 70 hours
Fibrinogen in mol/l | After 22 hours, 46 hours and 70 hours
Antithrombin in 10^3 int.units/l | After 22 hours, 46 hours and 70 hours
D-dimer in mg/l FEU | After 22 hours, 46 hours and 70 hours
Trombine time in seconds | After 22 hours, 46 hours and 70 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anni Norgaard Jeppesen, MD, Principal Investigator — Research Center of Emergency Medicine and Department of Anesthesiology and Intensive Care Medicine
Locations (1):
- Dept of Anesthesiology and Intensive Care and Dept of Clinical Biochemistry, Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] Jeppesen AN, Duez C, Kirkegaard H, Grejs AM, Hvas AM. Fibrinolysis in Cardiac Arrest Patients Treated with Hypothermia. Ther Hypothermia Temp Manag. 2023 Sep;13(3):112-119. doi: 10.1089/ther.2022.0037. Epub 2022 Dec 6. PMID 36473198
- [Derived] Jeppesen AN, Hvas AM, Duez CHV, Grejs AM, Ilkjaer S, Kirkegaard H. Prolonged targeted temperature management compromises thrombin generation: A randomised clinical trial. Resuscitation. 2017 Sep;118:126-132. doi: 10.1016/j.resuscitation.2017.06.004. Epub 2017 Jun 7. PMID 28602694